CLINICAL TRIAL: NCT05832450
Title: Validation of a Predictive Model to Calculate the Risk of Red Blood Cells Concentrates Transfusion in Patients Undergoing Elective Brain Tumours Resections
Brief Title: Predictive Model to Calculate the Risk of RBC Transfusion in Elective Brain Tumours Resections (TScoreBTR)
Acronym: TScoreBTR
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Hospital Clinic of Barcelona (Other); University of Salamanca (Other); Hospital de Leon (Other Government); Parc Taulí Hospital Universitari (Other); Hospital de Cruces (Other); Hospital del Mar (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Universitario Central de Asturias (Other); Hospital Son Espases (Other); Hospital Universitario Virgen de la Arrixaca (Other); Hospital General Universitario de Valencia (Other); Hospital Universitari de Bellvitge (Other); Hospital Miguel Servet (Other)
Responsible Party: Sponsor
Other Study IDs: TScoreBTR
Record Dates: First submitted 2022-12-09; First posted 2023-04-27 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Brain Tumor Adult; Transfusion; Surgery
Keywords: Predictive model; Risk of red blood cells concentrates transfusion; Brain tumours resections (primary or metastatic)
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- No intervention: Perioperative data of patient undergoing elective brain tumor resection without requirements of red cell concentrate transfusion.
  Interventions: Other: Red cell concentrate transfusion

INTERVENTIONS:
Other: Red cell concentrate transfusion — Perioperative data of patient undergoing elective brain tumor resection with requirements of red cell concentrate transfusion.

SUMMARY:
To validate a predictive model for the risk of receiving RBCs in this population. This model uses four preoperative values (haemoglobin levels, tumour volume, previous craniotomy in the same spot, and number of craniotomies foreseen). The investigators would like to create an online data collection tool and calculator.

DETAILED DESCRIPTION:
Observational study collecting data from different institutions and teams groups in Spain. The investigators aim at validating one model (published in Journal of Neurosurgical Anesthesiology) in different settings and populations to see if it can be accurately used to provide an opportunity to optimize both the patient and the surgical plan as well as to guide perioperative crossmatch and RBC orders.

Inclusion criteria - Brain tumour (primary or metastatic) patients undergoing craniotomy for resection.

Exclusion criteria Patients younger than 18 years old. Urgent/emergent surgery. Brain tumours not requiring full craniotomy. Patients with blood conditions causing coagulation abnormalities. Systemic disease associated with significant abnormalities in coagulation times (prothrombin time <60% or activated thromboplastin time > 50 sg).

Outcome The investigators aim at developing objective and simple criteria about the probability of requirements RBCs during a brain tumour resection surgery. This way we could create a simple tool that would help to optimize both the patient and the surgical plan as well as to guide perioperative crossmatch and RBCs orders.

Statistical Analysis

Transfusion requirement predictive probability will be calculated as follows:

〖1/(1+e〗^(-(5.7606 + [-0.7037*(PH in g/dL)+ 0.0103*(BTLTV in mm3)+ 1.0558*(NC)+ 0.6232*(PC)]))) PH: Preoperative haemoglobin; BTLTV: brain tumour lesions total volume; NC: craniotomies number; PC: previous craniotomy. NT=1 if NT>1, or 0; PC=1 if PC at the same site for resection (not only biopsy), or 0. Model discrimination and calibration will be assessed with area under ROC curve, and Hosmer-Lemeshow test with calibration plot, respectively. P<0.05 will indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

- Brain tumour (primary or metastatic) patients undergoing craniotomy for resection.

Exclusion Criteria:

* Patients younger than 18 years old.
* Urgent/emergent surgery.
* Brain tumours not requiring full craniotomy.
* Patients with blood conditions causing coagulation abnormalities.
* Systemic disease associated with significant abnormalities in coagulation times (prothrombin time <60% or activated thromboplastin time > 50 sg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing craniotomy for elective brain tumour resection (primary or metastatic).
Sampling Method: Probability Sample
Enrollment: 1434 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Number of red cell concentrate transfused | During the surgery
  Number of red cell concentrate transfused
Number of red cell concentrate transfused | Immediately (first 24 hours) after the surgery
  Number of red cell concentrate transfused

SECONDARY OUTCOMES:
Concentration of hemoglobine | Pre-surgery
  Concentration of pre-surgery hemoglobine
Brain tumor volume | Pre-surgery
  Brain tumor volume (mm3) on preoperative MRI
Number of patients with previous tumor craniotomy | Pre-surgery
  Number of patients with previous tumor craniotomy at the same place
Number of craniotomies | During the surgery
  Number of craniotomies

CONTACTS AND LOCATIONS:
Overall Officials: Martinez-Simon Antonio, PhD, MD, Principal Investigator — Department of Perioperative Medicine and Intensive Care
Locations (1):
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Tomas-Biosca A, Martinez-Simon A, Guridi J, Honorato-Cia C, Cacho-Asenjo E, Tejada Solis S, Bejarano B, Becerra-Castro MV, Nunez-Cordoba JM. Development and Performance Evaluation of a Clinical Predictive Model to Estimate the Risk of Red Blood Cell Requirements in Brain Tumor Surgery. J Neurosurg Anesthesiol. 2023 Jan 1;35(1):74-79. doi: 10.1097/ANA.0000000000000793. Epub 2021 Aug 16. PMID 34393176
- [Background] Tomas-Biosca A, Martinez-Simon A, Guridi J, Tejada Solis S, Bejarano B, Honorato-Cia C, Cacho-Asenjo E, Nunez-Cordoba JM. Preoperative Hemoglobin and Actual Need for Blood Transfusion in Brain Tumor Resection Procedures: A Retrospective Cohort Study. J Neurosurg Anesthesiol. 2022 Apr 1;34(2):251-252. doi: 10.1097/ANA.0000000000000753. No abstract available. PMID 33470594
- [Derived] Contreras-Lopez L, Clavero FI, Hurtado Restrepo PA, de Arriba NP, Alvarez AD, Montes Armenteros JA, Pellicena MP, Colorado AF, Asensi PD, Candil JF, Garcia LG, Albamonte PS, Krauchi OR, Nunez-Cordoba JM, Martinez-Simon A. Efficiency in packed red blood management for brain tumor resection: multicenter prospective cohort study (TScoreBTR). Blood Transfus. 2026 Jan-Feb;24(1):56-64. doi: 10.2450/BloodTransfus.1069. Epub 2025 Aug 28. PMID 40901795